CLINICAL TRIAL: NCT02064010
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Efficacy, Safety, and Pharmacokinetic Behavior of Orally Administered SNC-102 in Subjects With Drug-Induced Tardive Dyskinesia
Brief Title: A Phase 2 Trial Evaluating SNC-102 in Drug-Induced Tardive Dyskinesia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding terminated; company closed
Sponsor: Synchroneuron Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNC102-201
Record Dates: First submitted 2013-12-06; First posted 2014-02-17 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2016-11

CONDITIONS: Drug-induced Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — Acamprosate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SNC-102, low dose (Experimental): SNC-102 (Acamprosate calcium) tablet 4 week duration dosing
  Interventions: Drug: SNC-102
- SNC-102, high dose (Experimental): SNC-102 (Acamprosate calcium) tablet 4 week duration dosing
  Interventions: Drug: SNC-102
- Placebo (Placebo Comparator): Placebo tablet 4 week duration dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SNC-102 — Acamprosate calcium (SNC-102) tablet, administered orally for 4 weeks
  Other Names: Acamprosate calcium; Acamprosate calcium controlled-release tablet; calcium N-acetylhomotaurinate
  Arms: SNC-102, high dose; SNC-102, low dose
Drug: Placebo — Placebo tablet, administered orally for 4 weeks
  Arms: Placebo

SUMMARY:
This Phase 2 study was designed to evaluate the efficacy and safety of SNC-102 in subjects with drug-induced Tardive Dyskinesia (TD). To ensure an adequate evaluation of SNC-102, a randomized, double-blind, parallel-group, placebo-controlled trial was designed. Two dosing levels of SNC-102 are employed to evaluate the proposed dosing range. A target enrollment of 90 subjects with drug-induced TD will provide sufficient data to assess the efficacy and safety profiles of SNC-102 in the target population.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18-75 years of age.
2. Diagnosis, at least 3 months prior to the Screening Visit, of drug-induced TD

   1. AIMS ≥3 (moderate or worse) for ≥1 body area, or AIMS = 2 (mild) for ≥2 body areas; and
   2. >3 months exposure to antipsychotic drug or metoclopramide; and
   3. Other causes of dyskinesia have been ruled out.
3. AIMS score is confirmed at the Screening Visit by the Principal Investigator and the Trial Reading Center, and at the Baseline Visit at least 1 week later by the Principal Investigator.
4. If using antipsychotic medication or metoclopramide, dose has been stable for at least 60 days prior to the Baseline Visit and is expected to remain stable through the course of the trial.
5. If using opioid medication, dose has been stable for at least 14 days prior to the Baseline Visit and is expected to remain stable through the course of the trial.
6. If using vitamin or dietary supplements, dose and type has been stable for at least 14 days prior to the Baseline Visit and is expected to remain stable through the course of the trial.
7. If using alcohol, willingness to limit intake to no more than 2 drinks/day through the course of participation in the trial, and to abstain for at least 12 hours prior to any assessment visit.

Exclusion Criteria:

1. Unstable psychiatric status, as indicated by any change in psychotropic medication (unless approved by the Sponsor), or by hospitalization, within 60 days prior to the Screening Visit.
2. Active drug or alcohol dependence or abuse.
3. Current use of cocaine, amphetamine, phencyclidine (PCP), or ketamine, documented either by history or by urinary drug screening at Screening and Baseline Visits. Drugs used to treat attention deficit-hyperactivity disorder are allowed if stable for at least 14 days prior to the Baseline Visit and are expected to remain stable through the course of the trial.
4. Risk of significant medication non-adherence, based on the judgment of the Principal Investigator.
5. Neurologic or psychiatric disorder that could interfere with the attribution of observed involuntary movements to TD, such as a primary movement disorder unrelated to medication.
6. History of neuroleptic malignant syndrome.
7. Significant risk, in the judgment of the Principal Investigator, of suicidal or violent behavior.
8. Receipt of new medication for the treatment of TD within 4 weeks prior to the Baseline Visit or anticipated while participating in the trial.
9. Initiation of oral contraceptive medication, or change in dose, within 30 days prior to the Screening Visit, or anticipated while participating in the trial.
10. Gastrointestinal disease such as short-bowel or other malabsorption syndrome which, in the judgment of the Principal Investigator, could interfere with absorption of orally-administered medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by changes from baseline in summary scores on the Abnormal Involuntary Movement Scale (AIMS) | 4 weeks
  Determine the efficacy relative to placebo of SNC-102 in subjects with drug-induced tardive dyskinesia (TD), as assessed by changes from baseline to four weeks in summary scores on the Abnormal Involuntary Movement Scale (AIMS)

SECONDARY OUTCOMES:
Compare the effectiveness of low dose and high dose of SNC-102 | 4 weeks
  Compare the effectiveness of low dose and high dose, as assessed by changes from baseline to four weeks in summary scores on the Abnormal Involuntary Movement Scale (AIMS)
Assess safety and tolerability of SNC-102 in the tardive dyskinesia population | 4 weeks
  Nature and frequency of adverse events; changes from baseline in tests of psychiatric symptoms and cognitive function.
Assess the pharmacokinetic (PK) profile in TD subjects | 4 weeks
  Measure and analyze the serum concentration of acamprosate.
Determine the relationship between the PK profile and clinical effects of SNC-102 | 4 weeks
  Describe the correlation between change in AIMS score and serum levels of acamprosate.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA - Greater Los Angeles, Los Angeles, California, United States